CLINICAL TRIAL: NCT03863353
Title: Scenario Tailored Opioid Messaging Program (STOMP) to Improve Risk Understanding in Young Adults
Acronym: STOMPYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Terri Voepel-Lewis, Prinicipal Investigator, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: HUM00147378; 1R01DA044245-01A1 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-03-05 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pain, Postoperative; Medication Adherence; Opioid Use; Knowledge, Attitudes, Practice; Risk Reduction Behavior
MeSH Terms: conditions — Pain, Postoperative; Medication Adherence; Behavior; Risk Reduction Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: randomized, controlled, factorial design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Group assignment will be coded for subjects and data collectors. Subjects will be blinded to whether the information they receive is the Intervention vs. Control.
  Group assignment will coded on data entry and unblinded after analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Intervention (Experimental): This group will receive the scenario-tailored STOMP educational feedback
  Interventions: Behavioral: Educational Intervention
- Control (No Intervention): This group will receive only standard of care information.

INTERVENTIONS:
Behavioral: Educational Intervention — This intervention provides scenario-tailored opioid risk message feedback immediately following interactive analgesic decision-making exercises.
  Other Names: STOMP Intervention
  Arms: Education Intervention

SUMMARY:
Legitimate prescription opioid use during adolescence has been associated with later prescription opioid misuse and substance use disorder symptoms during adulthood. Thus, primary prevention interventions for older adolescents and young adults (15-24 yrs) at the time of prescribing are imperative.

The goal of our research is to improve opioid analgesic safety and efficacy by optimizing opioid risk recognition and informed decision-making among 15-24 year olds who are prescribed these agents for home use. Young adults and older adolescents who manage their own prescription pain medicines need to recognize opioid-related risks and make decisions that will both reduce these risks yet ensure effective pain relief. The proposed research will evaluate new strategies to help subjects learn about opioid risks and make safe and effective analgesic decisions. 355 subjects who are undergoing an elective surgical procedure will be recruited. Subjects will be randomized to receive the new educational routine information. Subjects' knowledge and perceptions will be evaluated at baseline and at critical times after surgery.

DETAILED DESCRIPTION:
The goal of this research is to improve opioid analgesic safety and efficacy by optimizing opioid risk recognition, informed decision-making including misuse among 15-24 year olds who are prescribed these agents for home use.

This is a randomized, controlled study design. The investigators will enroll emerging adults (aged 15-24 yrs) who are scheduled to undergo a surgical procedure and will be prescribed an opioid as part of their routine postoperative care. Comprehensive informed consent will be obtained.

No medical treatments will be altered for the purposes of this educational study. All participants will complete baseline surveys to assess their pain medicine familiarity, their opioid risk knowledge and perceptions, and their analgesic self-efficacy and their pain relief/ risk avoidance preferences. Participants will also be presented (via the survey platform) with several hypothetical (mock) scenarios and will be asked to make hypothetical decisions about how they would treat pain for each.

The Intervention group will receive tailored feedback and guidance after each scenario (i.e., the Scenario Tailored Opioid Messages) and the Control group will receive only routine analgesic risk and benefit information. Participants will complete the post-scenario/feedback surveys to re-assess opioid risk perceptions and self-efficacy and will complete brief health literacy surveys.

On days 7, 14 and at 1 and 3 months, participants will be resurveyed (via emailed qualtrics survey link or paper -whichever is preferred) about their opioid risk knowledge, perceptions, scenario decision making, analgesic self-efficacy and pain relief/risk avoidance preferences.

All surveys and datasheets will contain unique identifiers only. Identifiers will be maintained separately from survey data (linked only by unique identifier) to maintain privacy. Participants will receive up to $50 for participation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an elective surgical procedure for which it is expected they will receive a prescription pain medicine for management of pain during recovery at home.

Exclusion Criteria:

* Undergoing non-elective procedure
* Cognitive impairment precluding self-reporting of pain
* Hematologic/oncologic condition
* Liver of kidney conditions precluding usual analgesic prescription patters (opioid plus a non-opioid)
* Use of opioids for prolonged pain pre-operatively (<2 weeks)

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 503 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri Voepel-Lewis, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from 11/2019 through May 2021 from surgical clinic rosters at University of Michigan
Pre-assignment Details: Enrollment number includes all who "Started" by signing the consent and were assigned to study groups. "Completed" indicates those who were analyzed. "Not completed includes those withdrawn after signing consent but prior to analyses. Reasons incomplete are indicated below (reasons included; alterations in surgical procedure or no opioid prescription dispensed).
Period: Overall Study
Arm/Group | Education Intervention | Control
Started | 282 | 221
Completed | 258 | 201
Not Completed | 24 | 20
Not completed — incomplete baseline; surgical complication; no opioid prescription | 24 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Intervention | Control | Total
Number analyzed (Participants) | 258 | 201 | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (2.7) | 19.1 (2.8) | 19.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 104 | 238
  Male | 124 | 97 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 23
  Not Hispanic or Latino | 242 | 194 | 436
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 16 | 15 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 13 | 35
  White | 207 | 163 | 370
  More than one race | 11 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Opioid Risk Perception
Description: Perceived riskiness of opioid misuse (0-40 where 40 indicates highest risk perception)
Time Frame: Baseline, day 14, 3 months post intervention
Population: All who completed at least one follow-up measurement of risk perception.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 258 | 201
score on a scale
  Baseline | 31.4 (0.85) | 31.1 (1.01)
  Day 14 | 32.8 (.65) | 30.02 (1.12)
  Month 3 | 31.0 (.62) | 29.8 (1.21)
Statistical Analysis 1: Comparison: Education Intervention vs Control; Hypothesis was tested using multivariable regression models (generalized estimating equation); Test type: Superiority; p = .001, Regression, Linear — Adjusted for repeated measures and effects of covariates; Rebression coefficient = 2.13, 95% CI 2-sided [0.86 to 3.40]

2. Secondary Outcome: Opioid Misuse Intention Decisions
Description: Number of participants with opioid misuse intentions and behaviors
Time Frame: 3 months post intervention
Population: Rest of the sample lost to follow-up at months 1-3
Measure: Count of Participants; unit: Participants
Arm/Group | Education Intervention | Control
Number analyzed (Participants) | 226 | 173
Participants
  Misuse Intentions | 47 | 38
  Misuse behavior | 18 | 12
Statistical Analysis 1: Comparison: Education Intervention vs Control; Logistic regression model examined the effect of the intervention on the outcome (collapsed intentions/behaviors); Test type: Superiority; p = 0.534, Regression, Logistic — adjusted for covariates; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.72 to 1.90]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Review of medical records, clinic visits etc.
Arm/Group | Education Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/258 | 0/201
Serious Adverse Events (participants affected / at risk) | 9/258 | 6/201
Other Adverse Events (participants affected / at risk) | 0/258 | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Education Intervention (N=258) | Control (N=201)
Hospitalization (Surgical and medical procedures) | 9 (9) | 6 (6) — Unexpected hospitalizations or return to emergency room

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03863353/Prot_SAP_ICF_000.pdf